CLINICAL TRIAL: NCT02387970
Title: Non-inferiority Study of Immediate or Delayed Provisionalization at Posterior Healed Sites Using NobelParallelCC Implants
Brief Title: Immediate or Delayed Provisionalization in Posterior Healed Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Panos Papapanou, Professor of Dental Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAO5901
Record Dates: First submitted 2015-02-27; First posted 2015-03-13 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Partial Edentulism
Keywords: Dental implants; Partial edentulism; Immediate/delayed provisionalization
MeSH Terms: interventions — Crowns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate provisionalization (Active Comparator): Individuals will receive temporary dental crowns supported by NobelParallel CC implant at the same day as implant surgery
  Interventions: Procedure: Immediate provisionalization; Device: NobelParallel CC implant; Device: Dental crown
- Delayed provisionalization (Active Comparator): Individuals will receive temporary dental crowns supported by NobelParallel CC implant 3 months after implant surgery
  Interventions: Procedure: Delayed provisionalization; Device: NobelParallel CC implant; Device: Dental crown

INTERVENTIONS:
Procedure: Immediate provisionalization — Stage one protocol: Individuals will receive temporary crowns at the same day as implant surgery, and a final restoration at four months after surgery.
  Arms: Immediate provisionalization
Procedure: Delayed provisionalization — Stage two protocol: Individuals will receive temporary crowns 3 months after implant surgery, and a final restoration at four months after surgery.
  Arms: Delayed provisionalization
Device: NobelParallel CC implant — Supports the comprehensive range of dental prosthetics as well as full range of prefabricated abutments.
  Other Names: NobelParallel Conical Connection implant
Device: Dental crown — A tooth-shaped "cap" that is placed over a tooth or implant for teeth restoration and improvement in appearance.
  Other Names: Dental prosthetics

SUMMARY:
In this study, the investigators will examine the performance of a new dental implant that has been approved by the Food and Drug Administration for use to replace of missing teeth. The investigators will study two groups of patients: one group will receive a temporary crown to replace the missing tooth at the same day as implant surgery; the second group will receive a similar crown 3 months later. Both groups will receive a permanent crown on the implant 4 months after surgery, and will be followed up for a period of 12 months. The investigators want to examine whether the healing of the bone and gums surrounding the implant that receives a crown immediately is similar to the healing of the implant when the crown is delivered later. If this is indeed the case, then the investigators will be able to recommend faster treatment for all patients.

DETAILED DESCRIPTION:
Dental implants are a widely used treatment option for the replacement of lost teeth due to trauma or oral diseases. The original protocol for placement of dental implants in edentulous spaces in the maxilla or the mandible was introduced more than thirty years ago and called for a two-stage approach, i.e., surgical placement of submerged dental implants and subsequent uncovering with abutment connection, prosthesis fabrication and functional loading approximately 6 months after. Today, the time between surgery and loading in a two-stage protocol has been commonly abbreviated to 3-4 months, while immediate implant provisionalization has emerged as a reliable and predictable option in cases of adequate osseous support, having similar survival and success rates to the two-step procedure. Comparison of histological healing has demonstrated no significant differences in bone to implant contact between implants surgically placed according to a two-stage protocol and those immediately provisionalized. However, substantial variability was noted among the clinical protocols used in the studies carried out so far, and additional well-designed randomized controlled trials (RCTs) are needed to fully appreciate the clinical outcomes of immediate and early loading protocols.

The design of dental implants is a subject of continuous improvement, and implant manufacturers regularly introduce new products the use of which may result in accelerated soft and hard tissue healing, increased initial implant stability, and enhanced aesthetic outcomes. The purpose of this randomized, controlled trial is to compare treatment outcomes when using a newly-introduced dental implant (NobelParallel™ CC) in a one-stage or a two-stage protocol. This new implant has the same titanium oxide surface coating (TiUnite®) and the same design principles of the parallel-walled NobelSpeedy Groovy™ implants, and an internal conical connection. The implant is marketed under the premarket notifications K050406 and K073142 (510(k), Food and Drug Administration).

ELIGIBILITY:
Inclusion Criteria:

* 50 subjects will be recruited among those referred to the Columbia University College of Dental Medicine for tooth replacement using a dental implant in a posterior maxillary or mandibular region (premolar/molar area)
* Age 18 or older
* Healed extraction sockets (extraction carried out at least 3 months prior to recruitment)
* Implant site free of infection
* Systemically healthy patients or with controlled common systemic conditions
* Adjacent teeth present both mesially and distally to the implant site

Exclusion Criteria:

* Pregnancy or intent to be pregnant over the next 12 months
* Current smoking exceeding 10 cigarettes/day
* Parafunctional habits/ excessive occlusal forces
* Current orthodontic therapy
* Uncontrolled hypertension (blood pressure over 160/100) or poorly-controlled diabetes (HbA1c>8%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panos N Papapanou, DDS, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Dental Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branemark PI, Adell R, Albrektsson T, Lekholm U, Lundkvist S, Rockler B. Osseointegrated titanium fixtures in the treatment of edentulousness. Biomaterials. 1983 Jan;4(1):25-8. doi: 10.1016/0142-9612(83)90065-0. PMID 6838955
- [Background] Esposito M, Grusovin MG, Chew YS, Coulthard P, Worthington HV. One-stage versus two-stage implant placement. A Cochrane systematic review of randomised controlled clinical trials. Eur J Oral Implantol. 2009 Summer;2(2):91-9. PMID 20467608
- [Background] Piattelli A, Ruggeri A, Franchi M, Romasco N, Trisi P. An histologic and histomorphometric study of bone reactions to unloaded and loaded non-submerged single implants in monkeys: a pilot study. J Oral Implantol. 1993;19(4):314-20. PMID 8007025
- [Derived] Wang J, Lerman G, Bittner N, Fan W, Lalla E, Papapanou PN. Immediate versus delayed temporization at posterior single implant sites: A randomized controlled trial. J Clin Periodontol. 2020 Oct;47(10):1281-1291. doi: 10.1111/jcpe.13354. Epub 2020 Sep 4. PMID 32757387

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Started | 27 | 25
Completed | 26 | 23
Not Completed | 1 | 2
Not completed — Did not complete 1-year follow up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Provisionalization | Delayed Provisionalization | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Continuous [Mean (Full Range); unit: years] | 45.1 [25 to 63] | 48.8 [31 to 70] | 46.8 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 7 | 6 | 13
Tooth Type [Count of Participants; unit: Participants]
  Premolar | 12 | 9 | 21
  Molar | 14 | 14 | 28
Arch [Count of Participants; unit: Participants]
  Maxilla | 14 | 13 | 27
  Mandible | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Bone Level Mesial to the Implant
Description: Radiographic measurements of alveolar bone level mesial to the implant (at surgical placement and 6 months) will be carried out using the MIPACS software. The implant platform will be the reference point.
Time Frame: Baseline and 6 months
Population: Only includes individuals with analyzable data.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Number analyzed (Participants) | 24 | 21
Millimeters | 1.26 (1.10) | 1.85 (1.16)
Statistical Analysis 1: Comparison: Delayed Provisionalization; Test type: Superiority; p = 0.088, t-test, 2 sided

2. Primary Outcome: Radiographic Bone Level Mesial to the Implant
Description: Radiographic measurements of alveolar bone level mesial to the implant (at surgical placement and 12 months) will be carried out using the MIPACS software. The implant platform will be the reference point.
Time Frame: Baseline and 12 months
Population: Only includes individuals who completed the 1-year follow up.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Number analyzed (Participants) | 25 | 21
Millimeters | 1.14 (1.20) | 1.57 (1.17)
Statistical Analysis 1: Comparison: Delayed Provisionalization; Test type: Superiority; p = 0.235, t-test, 2 sided

3. Primary Outcome: Radiographic Bone Level Distal to the Implant
Description: Radiographic measurements of alveolar bone level distal to the implant (at surgical placement and 6 months) will be carried out using the MIPACS software. The implant platform will be the reference point.
Time Frame: Baseline and 6 months
Population: Only includes individuals with analyzable data.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Number analyzed (Participants) | 22 | 20
Millimeters | 1.36 (1.27) | 1.82 (0.76)
Statistical Analysis 1: Comparison: Delayed Provisionalization; Test type: Superiority; p = 0.165, t-test, 2 sided

4. Primary Outcome: Radiographic Bone Level Distal to the Implant
Description: Radiographic measurements of alveolar bone level distal to the implant (at surgical placement and 12 months) will be carried out using the MIPACS software. The implant platform will be the reference point.
Time Frame: Baseline and 12 months
Population: Only includes individuals who completed the 1-year follow up.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Number analyzed (Participants) | 23 | 21
Millimeters | 1.22 (1.40) | 1.60 (0.88)
Statistical Analysis 1: Comparison: Delayed Provisionalization; Test type: Superiority; p = 0.297, t-test, 2 sided

5. Secondary Outcome: Mean Change in Peri-implant Mucosal Margin Level
Description: Measurements of peri-implant mucosal margin levels will be measured at baseline and 6 months post-procedure.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: millimeters of tissue
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Number analyzed (Participants) | 22 | 17
millimeters of tissue | 0.28 (0.96) | -0.10 (0.65)
Statistical Analysis 1: Comparison: Delayed Provisionalization; Test type: Superiority; p = 0.121, t-test, 2 sided

6. Secondary Outcome: Mean Change in Peri-implant Mucosal Margin Level
Description: Measurements of peri-implant mucosal margin levels will be measured at baseline and 12 months post-procedure.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Number analyzed (Participants) | 21 | 16
millimeters | 0.27 (0.80) | -0.20 (0.92)
Statistical Analysis 1: Comparison: Delayed Provisionalization; Test type: Superiority; p = 0.248, t-test, 2 sided

7. Secondary Outcome: Mean Change in Peri-implant Mucosal Margin Level
Description: Measurements of peri-implant mucosal margin levels will be measured at 6 months and 12 months post-procedure.
Time Frame: 6 months and 12 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
Number analyzed (Participants) | 23 | 20
millimeters | 0.10 (0.76) | -0.08 (0.67)
Statistical Analysis 1: Comparison: Delayed Provisionalization; Test type: Superiority; p = 0.854, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 36 months from procedure
Arm/Group | Immediate Provisionalization | Delayed Provisionalization
All-Cause Mortality (participants affected / at risk) | 4/26 | 3/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 4/26 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Provisionalization (N=26) | Delayed Provisionalization (N=23)
Prosthetic Screw Loosening - Multiple (Product Issues) | 1 (1) | 2 (2)
Crown fracture (Product Issues) | 1 (1) | 0 (0) — Occurred 17 months after crown delivery
Prosthetic Screw Loosening - Single (Product Issues) | 1 (1) | 0 (0) — Occurred 16 months after crown delivery
Implant mobile/removed (General disorders) | 0 (0) | 1 (1) — Occurred 9 months after crown delivery
Cement - retained due to angle correction (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT02387970/Prot_SAP_000.pdf